CLINICAL TRIAL: NCT02261012
Title: Examination of the Pathological Mechanism of the Complex Regional Pain Syndrome of the Upper Limb in Comparison to Patients With Painful Carpal Tunnel Syndrome and Healthy Subjects - an Explorative Clinical Study
Brief Title: Examination of the Pathophysiologic Mechanisms of CRPS by Using QST, CPM, RIC, and Heart Rate Variability QST
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Head of the Dep. of Pain Management, Ruhr University of Bochum
Other Study IDs: CRPS2014
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Complex Regional Pain Syndrome; Carpal Tunnel Syndrome; Neuralgia
MeSH Terms: conditions — Complex Regional Pain Syndromes; Carpal Tunnel Syndrome; Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 30 healthy probands: group without the condition of interest
- 30 CRPS patients: group with condition of interest
- 30 CTS patients: group with a different type of pain on the upper limbs

SUMMARY:
This study aims for a better understanding of the pathophysiological mechanisms of the complex regional pain syndrome (CRPS). This will be done by testing the quantitative sensory testing, the remote ischemic conditioning, the conditioned pain modulation (CPM) and the analysis of the heart-rate variability in patients with CRPS and a control-group. We hypothesize decreased conditioned pain modulation, less effects of remote ischemic conditioning and an affection of the heart-rate variability in patients with CPRS.

DETAILED DESCRIPTION:
CRPS is an illness which (seriously) affects patients in their daily life activity. The fact that the pathophysiological mechanisms are not well understood yet makes it hard to treat these patients in the right manner.

Possible patho-mechanisms might be microvascular changes and dysfunctions of the inhibitory descending pain system. Furthermore, recent studies showed that CRPS patients have macrovascular changes and a lower blood level of NO on the affected side. This indicates a NO mediated perfusion dysfunction.

Aim of this study is to examine the pathophysiological mechanism of CRPS in relation to healthy subjects and patients with a different type of pain syndrome (carpal tunnel syndrome) on the upper limb.

The investigators try to get a better understanding of the changes in the pain inhibitory system and micro- and macrocirculating blood-systems, as well as of the autonomic system of CRPS-patients.

ELIGIBILITY:
CRPS-patients

Inclusion Criteria:

* Unilateral pain on the upper limbs, based on a scintigraphic ensured CRPS (average pain in the last 4 weeks ≥ 3 in pain Detect)
* Pain history < 1 year

Exclusion criteria:

* Bilateral pain on the upper limbs
* Inadequate knowledge of the german language in speaking and writing
* Acute psychiatric sickness
* Polyneuropathy
* Any added neuropathic sickness on the not affected upper limb sight
* Intolerable pain during the testing
* Injuries within the tested areal
* Acute injuries on the hand
* Pregnancy
* Missing informed consent

CTS-patients

Inclusion Criteria:

* Unilateral pain on the upper limbs, based on a scintigraphic ensured CRPS (average pain in the last 4 weeks ≥ 3 in pain Detect)
* Pain history < 1 year

Exclusion criteria:

* Bilateral pain on the upper limbs
* Inadequate knowledge of the german language in speaking and writing
* Acute psychiatric sickness
* Polyneuropathy
* Any added neuropathic sickness on the not affected upper limb sight
* Intolerable pain during the testing
* Injuries within the tested areal
* Acute injuries on the hand
* Pregnancy
* Missing informed consent

Healthy subjects

Inclusion Criteria:

* Age > 18 years
* Written consent

Exclusion criteria:

* Inadequate knowledge of the german language in speaking and writing
* Current pain
* Pain within in the last 14 days
* Any serious internistic medicin
* Any chronic skin disease
* Any central neural sickness
* Polyneuropathy
* Peripheral nerve lesion within the testing areal
* Any radiculopathy with permanent pain (in the last 3 months)
* Any psychiatric sickness
* Migraine ( at least one attack in the last 24 h)
* Repeating headache (in the last 3 month on >5 days/month)
* Taking any analgesics in the last 14 days
* Taking triptans in the last 24 months
* Taking any psychotropic's in the last 3 months
* Any repeated taking of medication, including amber or different psychostimulants (excluding contraceptives)
* Taking of any prescription and non-prescription drugs (except contraceptives) in the last 7 days or 5 half-life periods(which is always longer) before including into the study
* Achilles reflex absent or within in the side-difference pathologic hypoactive or hyperactive
* pallaesthesia <5/8 (<4/8 at >60 years) on the internal malleolus on both sides
* abuse of alcohol or medications/drugs (corresponding to the DSM IV criteria)
* joining a medical study <30 days before inclusion into the current study
* jet lag, irregular work schedule, sleep deprivation within the last 3 days
* change of intestity during physical activity, e.g. beginning an activity in the last weeks before inclusion into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, CRPS-patients, CTS-patients
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
CPM effect | 60 seconds
  Conditioned Pain Modulation measured by the Heat-Cold-Pain Method
Remote Ischemic Conditioning | 45 minutes
  the perfusion increasing effect after RIC in all groups

CONTACTS AND LOCATIONS:
Overall Officials: Tina Mainka, Dr. med., Principal Investigator — University Hospital Bergmannsheil, Department of Pain Medicine
Locations (1):
- Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil GmbH, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Hegelmaier T, Kumowski N, Mainka T, Vollert J, Goertz O, Lehnhardt M, Zahn PK, Maier C, Kolbenschlag J. Remote ischaemic conditioning decreases blood flow and improves oxygen extraction in patients with early complex regional pain syndrome. Eur J Pain. 2017 Sep;21(8):1346-1354. doi: 10.1002/ejp.1033. Epub 2017 Mar 24. PMID 28340289